CLINICAL TRIAL: NCT04860830
Title: A Phase III Randomized, Double-blind, Placebo-controlled Parallel Group Trial to Examine the Efficacy and Safety of Iclepertin Once Daily Over 26 Week Treatment Period in Patients With Schizophrenia (CONNEX-3)
Brief Title: CONNEX-3: A Study to Test Whether Iclepertin Improves Learning and Memory in People With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1346-0013; 2020-003726-23 (EudraCT Number)
Record Dates: First submitted 2021-04-26; First posted 2021-04-27 (Actual); Results first posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — BI 425809

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Iclepertin 10 mg (Experimental): Patients with schizophrenia took one tablet of 10 milligram (mg) iclepertin orally once daily for 26 weeks. Patients were permitted to remain on other antipsychotic and psychotropic medications, as specified in the eligibility criteria.
  Interventions: Drug: Iclepertin
- Placebo (Placebo Comparator): Patients with schizophrenia took one tablet of placebo matching iclepertin orally once daily for 26 weeks. Patients were permitted to remain on other antipsychotic and psychotropic medications, as specified in the eligibility criteria.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iclepertin — One tablet of 10 mg once daily for 26 weeks.
  Other Names: BI 425809
  Arms: Iclepertin 10 mg
Drug: Placebo — One tablet once daily for 26 weeks.
  Arms: Placebo

SUMMARY:
This study is open to adults with schizophrenia. Schizophrenia can affect the way a person thinks, their memory and their mental functioning. Examples include struggling to remember things, or to read a book or pay attention to a movie. Some people have difficulty calculating the right change or planning a trip so that they arrive on time. The purpose of this study is to find out whether a medicine called iclepertin improves learning and memory in people with schizophrenia.

Participants are put into two groups randomly, which means by chance. One group takes iclepertin tablets and the other group takes placebo tablets. Placebo tablets look like iclepertin tablets but do not contain any medicine. Participants take a tablet once a day for 26 weeks. In addition, all participants take their normal medication for schizophrenia.

During this time, doctors regularly test learning and memory of the participants by use of questionnaires, interviews, and computer tests. The results of the mental ability tests are compared between the groups.

Participants are in the study for about 8 months and visit the study site about 14 times. During this time, doctors regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria

* Signed and dated written informed consent.
* Male or female patients who are 18-50 years (inclusive) of age at time of consent.
* Diagnosis of schizophrenia utilizing Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5).

  -- Patients must be clinically stable and in the residual (non-acute) phase of their illness with no hospitalization or increase level of care due to worsening of schizophrenia in the past 12 weeks or no uncontrolled positive symptoms.
* Patients should have functional impairment in day-to-day activities per investigator judgement.
* Patients maintained on current antipsychotic treatment for at least 12 weeks and on current dose for at least 35 days prior to randomization.
* Patients with any other concomitant psychoactive medications (except for anticholinergics) need to be maintained on same drug for at least 12 weeks and on current dose/ regimen for at least 35 days prior to randomization.
* Women of childbearing potential must use highly effective methods of birth control.
* Have a study partner who interacts with the patient on a regular basis. Further inclusion criteria apply.

Exclusion criteria

* Patient with current DSM-5 diagnosis other than Schizophrenia.
* Cognitive impairment due to other causes, or patients with dementia or epilepsy.
* Severe movement disorders.
* Any suicidal behavior in past year or suicidal ideation in the past 3 months.
* History of moderate or severe substance use disorder within the last 12 months prior to informed consent.
* Positive urine drug screen.
* Patients who were treated with Clozapine, stimulants, ketamine or electroconvulsive therapy within 6 months prior to randomization.
* Current participation in any investigational drug trial.
* Cognitive Remediation Therapy within 12 weeks prior to screening.
* Initiation or change in any type or frequency of psychotherapy within 12 weeks prior to randomization.
* Any clinically significant finding or condition that would jeopardize the patient´s safety while participating in the trial or their capability to participate in the trial.
* Haemoglobin (Hb) below lower limit of normal .
* History of haemolytic anaemia, red blood cell (RBC) membrane diseases, known Glucose-6-phosphate dehydrogenase deficiency, anaemia of any cause or patients planning to donate blood.
* Severe renal impairment.
* Indication of liver disease.
* Any documented active or suspected malignancy or history of malignancy within 5 years.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.

Further exclusion criteria apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 609 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-11-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (110):
- United States (24):
  - Advanced Research Center, Inc., Anaheim, California
  - ProScience Research Group, Culver City, California
  - University of California Los Angeles, Los Angeles, California
  - CNRI - Los Angeles, Pico Rivera, California
  - Stanford University Medical Center, Stanford, California
  - Sunwise Clinical Research-Walnut Creek-70166, Walnut Creek, California
  - Advanced Medical Research Group Inc, Hollywood, Florida
  - Accel Research Sites Network, Maitland, Florida
  - University of Miami, Miami, Florida
  - Ivetmar Medical Group, LLC, Miami, Florida
  - Nova Psychiatry Inc., Orlando, Florida
  - Synexus Clinical Research-Atlanta-67262, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Center for Behavioral Health, LLC, Gaithersburg, Maryland
  - Arch Clinical Trials, LLC, St Louis, Missouri
  - Omaha Insomnia and Psychiatric Services, Omaha, Nebraska
  - Hassman Research Institute-Berlin-60540, Berlin, New Jersey
  - UNC Center for Excellence in Community Mental Health, North Carolina Psychiatric Research Center, Raleigh, North Carolina
  - Midwest Clinical Research, Dayton, Ohio
  - Rivus Wellness and Research Institute, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Oasis Life Care, State College, Pennsylvania
  - Ben Taub General Hospital, Houston, Texas
  - LinQ Research, LLC-Richmond-70076, Richmond, Texas
- Argentina (9):
  - Clínica Privada Banfield, Banfield
  - Fundación para el Estudio y Tratamiento de las Enfermedades Mentales (FETEM), CABA
  - Fundación FunDaMos para la asistencia e investigación en psiquiatría, CABA
  - CEN (Centro Especializado Neurociencias), Córdoba
  - Instituto Modelo de Neurología Lennox, Córdoba
  - Instituto Médico DAMIC S.R.L., Córdoba
  - Instituto de Neurociencias San Agustín, La Plata
  - Instituto Médico de la Fundación Estudios Clínicos, Rosario
  - Centro Medico Luquez, San Vicente
- AKH - Medical University of Vienna, Vienna, Austria
- Belgium (4):
  - CUP Vivalia -La Clairière, Bertix
  - Sint-Kamillus, Bierbeek
  - Universitair Psychiatrisch Centrum Duffel (UPC Duffel), Duffel
  - Meclinas, Mechelen
- Brazil (2):
  - Ruschel Medicina e Pesquisa Clínica, Rio de Janeiro
  - Clínica Viver - Centro de Desospitalização Humana, São Paulo
- Bulgaria (3):
  - Filipopolis Ambulatory for Group Practice for Specialized Care in Psychiatry, Plovdiv
  - Medical Center "Spectar", Plovdiv
  - Medical Center Hera EOOD, Sofia
- China (11):
  - Beijing Anding Hospital, Beijing
  - The Second Xiangya Hospital Of Central South University, Changsha
  - The third affiliated hospital of Sun Yat-Sen University, Guangzhou
  - Huzhou Third Municipal Hospital, Huzhou
  - Nanjing Brain Hospital, Nanjing
  - Shenzhen Kangning Hospital, Shenzhen
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - Tianjin Anding Hospital, Tianjin
  - First Affiliated Hospital of Xi'an JiaoTong University, Xi'an
  - Xi'an Mental Health Center, Xi'an
  - Zhumadian Psychiatric Hospital, Zhumadian
- Czechia (6):
  - National Institute of Mental Health, Klecany
  - MP Meditrine s.r.o., Ostrava
  - A-SHINE s.r.o, Pilsen
  - PRAGTIS s.r.o., Prague
  - INEP medical s.r.o., Prague
  - Psychiatrie Ricany s.r.o., Říčany
- Denmark (3):
  - Aalborg Universitetsshospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Psykiatrisk Center Glostrup, Glostrup Municipality
- Finland (3):
  - HUS Jorvi Hospital, Espoo
  - Aurora hospital, Helsinki
  - CRST - Clinical Research Services Turku, Turku
- Germany (5):
  - Studienzentrum für Neurologie und Psychiatrie, Böblingen
  - LWL-Klinik Dortmund, Dortmund
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Klinikum der Universität München - Campus Innenstadt, München
  - Universitätsklinikum Tübingen, Tübingen
- Lithuania (4):
  - JSC Romuvos Clinic, Kaunas
  - LUHS KH Psichiatric Clinic Mariu Division, Kaunas
  - JSC Medical center "Puriena", Šilutė
  - Vilnius City Mental Health Center, Vilnius
- Mexico (7):
  - Centro de Investigacion Integral MEDIVEST S.C, Chihuahua City
  - Centro para el Desarrollo de la Medicina y de Asistencia Medica Especializada S.C., Culiacán
  - Hospital Aranda de la Parra, León
  - Centro de Investigación Clinica Acelerada, S.C., Mexico City
  - Iecsi S.C., Monterrey
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
  - BIND Investigaciones S.C., San Luis Potosí City
- Portugal (3):
  - ULS da Região de Leiria, E.P.E., Leiria
  - ULS de Santa Maria, E.P.E, Lisbon
  - ULS de Loures-Odivelas, E.P.E, Loures
- Serbia (3):
  - Clinical Hospital Center Dr. Dragisa Misovic, Belgrade
  - General Hospital Euromedik, Belgrade
  - Special Hospital for Psychiatric Diseases Gornja Toponica, Gornja Toponica
- South Korea (6):
  - Inje University Busan Paik Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Seongnam
  - CHA Bundang Medical Center, Seongnam-si
  - Pusan National University Yangsan Hospital, Yangsan
- Taiwan (8):
  - Kai-Syuan Psychiatric Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital-Keelung, Keelung
  - Chung Shan Medical University Hospital, Taichung
  - NCKUH, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
  - Taoyuan Psychiatric Center, Taoyuan District
- United Kingdom (8):
  - Bodmin Community Hospital, Bodmin
  - The Fritchie Centre, Cheltenham
  - Redesmere, Chester
  - Western General Hospital, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow
  - Maudsley Hospital, London
  - Warneford Hospital, Oxford
  - Moorgreen Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Keefe RSE, Harvey PD, Correll CU, Falkai P, Hashimoto N, Klein H, Krystal JH, Marder S, Medalia A, Sumiyoshi T, Wang G, Zhang H, Blahova Z, Bichard-Sall I, English BA, Fu E, Gruenenfelder F, Groeschl M, Kimura K, Tang W, von der Goltz C, Fowler C. Efficacy and safety of iclepertin for cognitive impairment associated with schizophrenia (CONNEX programme): results from three phase 3 randomised controlled trials. Lancet Psychiatry. 2025 Dec;12(12):906-920. doi: 10.1016/S2215-0366(25)00296-2. PMID 41233083
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multi-center, multi-national, randomized, double-blind, placebo controlled, parallel group, 26-week trial in patients with schizophrenia on stable antipsychotic treatment randomized with equal ratio to iclepertin or placebo.
  Patients who completed the trial could directly enroll into a open-label extension trial to assess the long-term safety and tolerability of iclepertin (1346-0014). A dedicated ocular sub-study was conducted in several countries to investigate the ocular safety of iclepertin.
Pre-assignment Details: Patients and study partners signed informed consent forms and were informed that they were free to withdraw consent at any time without penalty or prejudice. All patients were screened for eligibility prior to participation and attended a specialist site which ensured that they strictly met all inclusion and no exclusion criteria. Study partners were not enrolled nor assigned a study ID, and other than the endpoints related to patients, no other data was collected from them.
Period: Overall Study
Arm/Group | Iclepertin 10 mg | Placebo
Started | 303 (This is the number of randomized patients.) | 306 (This is the number of randomized patients.)
Treated | 301 | 305
Ocular safety sub-study | 36 | 38
Completed | 271 | 258
Not Completed | 32 | 48
Not completed — Adverse Event | 8 | 18
Not completed — Perceived lack of efficacy | 1 | 6
Not completed — Change of residence | 4 | 2
Not completed — Burden of study procedures | 2 | 4
Not completed — No reason available | 3 | 2
Not completed — Subject decision | 9 | 12
Not completed — Physician Decision | 1 | 0
Not completed — Other than listed | 2 | 3
Not completed — Not treated | 1 | 0
Not completed — Randomized in error and not treated | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Set (RS): all patients who signed informed consent and were randomized into the trial, regardless of whether they were treated with trial medication. Patients randomized in error and discontinued from the study before the start of trial medication were excluded from the RS. Baseline characteristics were not collected for study partners.
Groups:
- Total: Total of all reporting groups
Arm/Group | Iclepertin 10 mg | Placebo | Total
Number analyzed (Participants) | 302 | 305 | 607
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.3 (8.7) | 33.4 (8.8) | 33.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 130 | 224
  Male | 208 | 175 | 383
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 71 | 83 | 154
  Not Hispanic or Latino | 231 | 222 | 453
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 7 | 17
  Asian | 112 | 116 | 228
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 27 | 24 | 51
  White | 149 | 155 | 304
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Overall composite T-score of the MATRICS consensus cognitive battery (MCCB) [Mean (Standard Deviation); unit: T-score] — The Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) consensus cognitive battery (MCCB) assesses 7 cognitive domains, including speed of processing, attention vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. T-scores in the general population have a mean of 50 and standard deviation of 10, and a higher score indicates better cognition.
  T-score | 29.4 (14.1) | 29.8 (13.5) | 29.6 (13.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Overall Composite T-score of the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) After 26 Weeks of Treatment
Description: The MCCB assesses 7 cognitive domains, including speed of processing, attention vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. T-scores in the general population have a mean of 50 and standard deviation of 10, and a higher score indicates better cognition. The primary analysis was a restricted maximum likelihood (REML) based approach using a mixed-effects model for repeated measurements (MMRM), which included the fixed categorical effects of treatment at each visit, fixed categorical effect of the stratification factor using the screening MCCB overall composite T-score, and a fixed effect for the continuous covariate of baseline at each visit. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-subject dependencies. Intercurrent events were addressed using different pre-defined strategies.
Time Frame: The MMRM model incorporates values from baseline (Week 0), Week 12 and Week 26. The data represent the Least Squares Means at Week 26.
Population: Randomized Set (RS): all patients who signed informed consent and were randomized into the trial, regardless of whether they were treated with trial medication. Patients randomized in error and discontinued from the study before the start of trial medication were excluded from the RS.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Iclepertin 10 mg | Placebo
Number analyzed (Participants) | 302 | 305
T-score | 1.890 (0.3336) | 2.273 (0.3372)
Statistical Analysis 1: Comparison: Iclepertin 10 mg vs Placebo; The primary analysis was a REML-based approach using a MMRM, which included the fixed categorical effects of treatment at each visit, fixed categorical effect of the stratification factor using the screening MCCB overall composite T-score, and a fixed effect for the continuous covariate of baseline at each visit. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-subject dependencies; Test type: Superiority; p = 0.4187, Mixed Models Analysis — Null hypothesis: the adjusted mean change in iclepertin is worse than or equal to that in placebo. One-sided significance level of <0.025 is needed for conducting further formal hypothesis tests in the secondary endpoints; Difference of adjusted means = -0.384, 95% CI 2-sided [-1.316 to 0.548], Standard Error of Mean 0.4745 — Adjusted mean iclepertin - adjusted mean placebo

2. Secondary Outcome: Change From Baseline in the Schizophrenia Cognition Rating Scale (SCoRS) Interviewer Total Score After 26 Weeks of Treatment
Description: SCoRS is a 20-item interview-based assessment of cognitive deficits and the degree to which they affect day-to-day functioning. Each item is rated on a 4-point scale. Higher ratings reflect a greater degree of impairment. The interviewer integrates information from separate patient and study partner interviews to generate a total score, which ranges from 20 to 80. The analysis was a REML-based approach using a MMRM model, which included the discrete fixed effects of treatment at each visit, fixed categorical covariate of the stratification factor using the screening MCCB overall composite T-score, a fixed effect for the continuous covariate of baseline at each visit. Visit was treated as the repeated measure with an unstructured covariance structure to model the within-subject measurements. Subjects were considered as a random effect. Intercurrent events were addressed using different pre-defined strategies.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Iclepertin 10 mg | Placebo
Number analyzed (Participants) | 302 | 305
Scores on a scale | -3.751 (0.3697) | -4.513 (0.3728)
Statistical Analysis 1: Comparison: Iclepertin 10 mg vs Placebo; The analysis was a REML-based approach using a MMRM model, which included the discrete fixed effects of treatment at each visit, fixed categorical covariate of the stratification factor using the screening MCCB overall composite T-score, a fixed effect for the continuous covariate of baseline at each visit. Visit was treated as the repeated measure with an unstructured covariance structure to model the within-subject measurements. Subjects were considered as a random effect; Test type: Other; p = 0.1478, Mixed Models Analysis; Difference of adjusted means = 0.762, 95% CI 2-sided [-0.271 to 1.794], Standard Error of Mean 0.5255 — Adjusted mean iclepertin - adjusted mean placebo

3. Secondary Outcome: Change From Baseline to Week 26 in the Adjusted Total Time T-score in Virtual Reality Functional Capacity Assessment Tool (VRFCAT)
Description: The VRFCAT is a virtual reality shopping trip performed on a tablet, and was used as an electronic Functional Capacity measure by measuring the total time adjusting for the number of errors. T-scores in the general population have a mean of 50 and standard deviation of 10, and a higher score indicates a better functional outcome. The analysis was a REML-based approach using a MMRM model, which included the discrete fixed effects of treatment at each visit, fixed categorical covariate of the stratification factor using the screening MCCB overall composite T-score, a fixed effect for the continuous covariate of baseline at each visit. Visit was treated as the repeated measure with an unstructured covariance structure to model the within-subject measurements. Subjects were considered as a random effect. Intercurrent events were addressed using different pre-defined strategies.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Iclepertin 10 mg | Placebo
Number analyzed (Participants) | 302 | 305
T-score | 1.820 (0.7633) | 3.042 (0.7669)
Statistical Analysis 1: Comparison: Iclepertin 10 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.2596, Mixed Models Analysis; Difference of adjusted means = -1.221, 95% CI 2-sided [-3.347 to 0.904], Standard Error of Mean 1.0820 — Adjusted mean iclepertin - adjusted mean placebo

4. Secondary Outcome: Change From Baseline to Week 26 in the T-score of the Number of Correct Responses on Tower of London
Description: This is an Executive Functions/Reasoning and Problem Solving test where patients were shown two images on opposite sides of a tablet screen. Each image showed a different configuration of 3 colored balls arranged on 3 pegs. Patients were required to accurately determine the total number of times the balls in one picture would have to be moved in order to make the arrangement of balls identical to that of the other opposing picture, while employing the standard rules employed in tower tests. T-scores in the general population have a mean of 50 and standard deviation of 10, and a higher score indicates a better outcome. The analysis was performed with an analysis of covariance (ANCOVA) model, which included treatment, stratification factor of screening MCCB overall composite T-score (< 30, ≥ 30), and baseline number of correct responses on Tower of London T-score.
Time Frame: At baseline (Week 0) and at Week 26.
Population: Randomized Set (RS): all patients who signed informed consent and were randomized into the trial, regardless of whether they were treated with trial medication. Patients randomized in error and discontinued from the study before the start of trial medication were excluded from the RS. Only patients with available data at Week 26 were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Iclepertin 10 mg | Placebo
Number analyzed (Participants) | 280 | 277
T-score | 0.440 (0.5773) | 1.016 (0.5805)
Statistical Analysis 1: Comparison: Iclepertin 10 mg vs Placebo; The analysis was performed with an ANCOVA model, which included treatment, stratification factor of screening MCCB overall composite T-score (< 30, ≥ 30), and baseline number of correct responses on Tower of London T-score; Test type: Other; p = 0.4822, ANCOVA; Difference of adjusted means = -0.576, 95% CI 2-sided [-2.184 to 1.032], Standard Error of Mean 0.8187 — Adjusted mean iclepertin - adjusted mean placebo

5. Secondary Outcome: Change From Screening Visit 1a to Week 24 in Patient Reported Experience of Cognitive Impairment in Schizophrenia (PRECIS) Total Score
Description: PRECIS consists of 26 items covering 6 domains (memory, communication, self-control, executive function, attention, and sharp thinking), and 2 additional items assessing the overall degree of bother associated with all domains. Questions are answered via a 5-category Likert scale, with higher scores indicating a worse patient experience. The total score, ranging from 26 to 130, is the average score of the first 26 items. The analysis was a REML-based approach using a MMRM model, which included the discrete fixed effects of treatment at each visit, fixed categorical covariate of the stratification factor using the screening MCCB overall composite T-score, and continuous fixed effects for the corresponding baseline endpoint value at each visit. Visit was treated as the repeated measure with an unstructured covariance structure to model the within-subject measurements. Subjects were considered as a random effect. Intercurrent events were addressed using different pre-defined strategies.
Time Frame: The MMRM model incorporates values from baseline (screening), Week 15 and Week 24. The data represent the Least Squares Means at Week 24.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Iclepertin 10 mg | Placebo
Number analyzed (Participants) | 302 | 305
Scores on a scale | -0.275 (0.0274) | -0.234 (0.0278)
Statistical Analysis 1: Comparison: Iclepertin 10 mg vs Placebo; The analysis was a REML-based approach using a MMRM model, which included the discrete fixed effects of treatment at each visit, fixed categorical covariate of the stratification factor using the screening MCCB overall composite T-score, and continuous fixed effects for the corresponding baseline endpoint value at each visit. Visit was treated as the repeated measure with an unstructured covariance structure to model the within-subject measurements. Subjects were considered as a random effect; Test type: Other; p = 0.2936, Mixed Models Analysis; Difference of adjusted means = -0.041, 95% CI 2-sided [-0.118 to 0.036], Standard Error of Mean 0.0391 — Adjusted mean iclepertin - adjusted mean placebo

6. Secondary Outcome: Ocular Safety Sub-study: Change From Baseline in Humphrey Visual Field 24-2 Swedish Interactive Thresholding Algorithm (SITA) Standard at Week 24
Description: The Humphrey visual field is a diagnostic test to measure visual fields, or perimetry. The Humphrey visual field test measures the entire area of peripheral vision that can be seen while the eye is focused on a central point. During this test, lights of varying intensities appear in different parts of the visual field while the patient's eye is focused on a central spot. The perception of these lights is charted and then compared to results of a healthy eye at the same age of the patient to determine if any damage has occurred. Visual field Index goes from 100%= perfect to 0= no vision.
Time Frame: Measurements were performed at baseline (screening) and at Week 24.
Population: Ocular sub-study Set (EYE): all treated patients who consented to participate in the ocular sub-study (including late/retrospective consent to the ocular sub-study) and had evaluable ophthalmologic measurements.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Iclepertin 10 mg | Placebo
Number analyzed (Participants) | 26 | 32
Units on a scale
  Left eye | 2.00 (6.06) | -3.97 (12.99)
  Right eye | -0.31 (3.56) | -4.44 (15.51)

7. Secondary Outcome: Ocular Safety Sub-study: Change From Baseline in Spectral Domain Ocular Coherence Tomography (OCT)
Description: The central retinal thickness measurements were recorded for each eye via high definition optical coherence tomography (spectral domain OCT) to evaluate the retinal and sub-retinal structures.
Time Frame: Measurements were performed at baseline (screening) and at Week 24.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Micrometer (µm)
Arm/Group | Iclepertin 10 mg | Placebo
Number analyzed (Participants) | 28 | 32
Micrometer (µm)
  Left eye | -1.57 (7.25) | -1.47 (10.08)
  Right eye | -1.14 (5.70) | -2.41 (11.75)

ADVERSE EVENTS:
Time Frame: From first treatment administration until last treatment administration plus residual effect period, up to approximately 31 weeks.
Description: Treated Set (TS): includes all patients who signed informed consent and were treated with at least one dose of the trial medication. Study partners were not assessed or monitored for deaths and adverse events.
Arm/Group | Iclepertin 10 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/301 | 0/305
Serious Adverse Events (participants affected / at risk) | 13/301 | 14/305
Other Adverse Events (participants affected / at risk) | 68/301 | 65/305
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iclepertin 10 mg (N=301) | Placebo (N=305)
Central serous chorioretinopathy (Eye disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 1
Schizophrenia (Psychiatric disorders) | 3 | 2
Suicidal behaviour (Psychiatric disorders) | 0 | 2
Suicidal ideation (Psychiatric disorders) | 3 | 6
Suicide attempt (Psychiatric disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Iclepertin 10 mg (N=301) | Placebo (N=305)
Nasopharyngitis (Infections and infestations) | 17 | 19
Weight increased (Investigations) | 11 | 20
Headache (Nervous system disorders) | 28 | 22
Schizophrenia (Psychiatric disorders) | 20 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT04860830/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-23): https://cdn.clinicaltrials.gov/large-docs/30/NCT04860830/SAP_001.pdf